CLINICAL TRIAL: NCT00741208
Title: Modification of Asthma With Soy Isoflavone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Respiratory Health Association of Metropolitan Chicago (Other)
Responsible Party: Ravi Kalhan, MD, MS, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 2804
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
Keywords: asthma; soy isoflavone; genistein; soy
MeSH Terms: conditions — Asthma | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Patients randomized to receive soy isoflavone twice daily for 2 weeks. Patients will cross-over and receive placebo medication for 2 weeks later in the study
  Interventions: Dietary Supplement: Soy Isoflavone
- 2 (Other): Patients randomized to receive placebo medication twice daily for 2 weeks. Patients will cross-over and receive soy isoflavone for 2 weeks later in the study
  Interventions: Dietary Supplement: Soy Isoflavone

INTERVENTIONS:
Dietary Supplement: Soy Isoflavone — 50mg soy isoflavone supplement consumed twice daily for a total of 100mg of soy isoflavones per day.

SUMMARY:
The purpose of this study is to determine if dietary supplementation with soy isoflavones in persistent asthma improves airway reactivity as determined by PC20 to methacholine.

DETAILED DESCRIPTION:
Asthma is a complex disease whose prevalence and severity are determined by multiple genetic and environmental factors. The prevalence of asthma has increased during the past few decades. Although causal relationships have not been proven, changing dietary practices have paralleled the increase in asthma prevalence. Several surveys have found an association between reduced lung function and decreased consumption of antioxidants, flavonoids, and essential vitamins in a variety of respiratory conditions including asthma. These findings suggest that diet may be a factor that impacts asthma and its clinical manifestations.

Higher dietary consumption of soy isoflavones is associated with decreased self-report of cough and other allergic respiratory symptoms. Our group reported an inverse relationship between dietary intake of the soy isoflavone genistein and asthma severity. In addition, we recently demonstrated that genistein inhibits synthesis of cysteinyl-leukotrienes in eosinophils by blocking p38-dependent activation of 5-lipoxygenase, providing a plausible cellular mechanism for the benefit of soy isoflavones in asthma. We also documented that dietary soy isoflavone supplementation in asthma patients inhibited eosinophil cysteinyl-leukotriene synthesis and decreased exhaled nitric oxide, an indicator of eosinophilic airway inflammation. Our overall long-term goal is to translate these epidemiological and mechanistic findings to human disease and determine whether dietary soy isoflavones have a clinical role in asthma. We propose a clinical study powered to detect an improvement in lung function as the first stop in achieving this goal.

Our hypothesis is that dietary supplementation with isoflavones will improve lung function, reduce symptoms, and decrease airway inflammation in asthma. To test this, we will conduct a randomized placebo-controlled, cross-over study of soy isoflavone supplementation in patients with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Physician diagnosed asthma;
* Positive methacholine bronchoprovocation test (20% fall in FEV1 at less than 8 mg/ml) with the past 3 years;
* Smoking Status: non-smoker for 6 months or longer and a less than 10 pack-year cumulative smoking history.

Exclusion Criteria:

* Pulmonary function FEV1< 70% predicted pre-bronchodilator;
* Other major chronic illness: conditions that in the judgement of athe principle investigator would interfere with participation in the study or history of or physician diagnosis of COPD, emphysema, or chronic bronchitis;
* Medication use: current consumption of soy isoflavone supplements or oral corticosteroid use within the past 6 months OR use of an investigational treatment within the previous 30 days;
* Drug allergy: known adverse reaction to genistein, other phytoestrogens, or soy products;
* Females of childbearing potential: pregnant or lactating or women of appropriate ago who report the possibility of pregnancy at the time of enrollment will be screened and cannot participate if pregnant;
* Non-adherence: inability or unwillingness to provide informed consent or inability to swallow study medication or inability to perform baseline measurements or completion of fewer than 5 of the 7 days of screening period diary entry or inability to be contacted by telephone;
* Other exclusions: recent asthma exacerbation (within 6 weeks) or recent upper respiratory tract infection (within 2 weeks) or change in diet over the past 1 month or expected change in diet (for example a weight loss diet) during the 6 week study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change in airway reactivity induced by dietary supplementation with soy isoflavones. Airway reactivity will be measured with methacholine bronchoprovocation testing. | 6 weeks

SECONDARY OUTCOMES:
Change in FEV1, morning peak flow rate, asthma control, markers of airway hyperreactivity and inflammation including sputum eosinophilia and eosinophilic cationic protein, fraction of expired nitric oxide, and urinary leukotriene. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Kalhan, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States